CLINICAL TRIAL: NCT05254158
Title: Investigation of Pharmacokinetic Properties of Single Subcutaneous Doses of NNC0174-0833 in Chinese Male Subjects Being Normal Weight, Overweight or With Obesity
Brief Title: A Research Study of How NNC0174-0833 Behaves in Chinese Volunteers Who Are Normal Weight, Overweight or With Obesity
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NN9838-4615; U1111-1247-7538 (Other: World Health Organization (WHO))
Record Dates: First submitted 2022-02-15; First posted 2022-02-24 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NNC0174 0833 1.8 mg (Experimental): Each participant will receive one single dose of NNC0174 0833
  Interventions: Drug: NNC0174 0833
- NNC0174 0833 0.9 mg (Experimental): Each participant will receive one single dose of NNC0174 0833
  Interventions: Drug: NNC0174 0833
- NNC0174 0833 0.3 mg (Experimental): Each participant will receive one single dose of NNC0174 0833
  Interventions: Drug: NNC0174 0833

INTERVENTIONS:
Drug: NNC0174 0833 — Participants will either get a single dose of 0.3 mg, 0.9 mg or 1.8 mg NNC0174-0833, administered subcutaneously (s.c., under the skin)

SUMMARY:
The aim of this study is to look at how the study medicine behaves in participants body and how it is removed from their body.

The study compares three different doses of the study medicine in Chinese healthy men.

Participant will either get 0.3 mg, 0.9 mg or 1.8 mg NNC0174-0833 which dose participant get is decided by chance.

NNC0174-0833 is a new medicine and has not been approved by the Center for Drug Evaluation.

We are testing the study medicine to make a medicine that can help people lose weight.

Participant will get 1 injection by a study nurse or doctor at the clinic. The injection will be with a needle in a skin fold in the stomach area.

The study will last for about 5 months. But participants participation will last about 2 months.

Participant will have 8 clinic visits with the study staff. One of these visits will be a 7-day, 6-night stay.

At all visits, except the information visit, participant will have blood drawn along with other clinical examinations.

Participants will be asked about their health, medical history and habits including mental health.

ELIGIBILITY:
Key inclusion criteria

* Chinese male subject aged 18-55 years (both inclusive) at the time of signing informed consent.
* Body mass index (BMI) between 20.0 and 39.9 kg/m^2 (both inclusive) at screening.
* Body weight between 60.0 and 110.0 kg (both inclusive) at screening.

Key exclusion criteria

* Male subject who is not sexually abstinent or surgically sterilised (vasectomy) or who or whose partner(s) is not willing to use highly effective contraceptive methods (as required by local regulation or practice) throughout the trial (until 'end of trial').
* Any disorder, which in the investigator's opinion might jeopardise subject's safety or compliance with the protocol.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
AUC0-∞, NNC0174-0833: The area under the NNC0174-0833 plasma concentration-time curve from time 0 to infinity after a single dose | From pre-dose (Day 1) to Visit 7 (Day 36)
  measured in h·nmol/L

SECONDARY OUTCOMES:
AUC0-168, NNC0174-0833: The area under the NNC0174-0833 plasma concentration-time curve from time 0 to 168 hours after a single dose | From pre-dose (Day 1) to Visit 3 (Day 8)
  measured in h·nmol/L
Cmax, NNC0174-0833: The maximum concentration of NNC0174-0833 in plasma | From pre-dose (Day 1) to Visit 7 (Day 36)
  measured in nmol/L
tmax, NNC0174-0833: The time from dose administration to maximum plasma concentration of NNC0174-0833 | From pre-dose (Day 1) to Visit 7 (Day 36)
  measured in hours
t1/2, NNC0174-0833: The terminal half-life of NNC0174-0833 | From pre-dose (Day 1) to Visit 7 (Day 36)
  measured in hours
CL/FNNC0174-0833: The apparent total plasma clearance of NNC0174-0833 | From pre-dose (Day 1) to Visit 7 (Day 36)
  measured in L/h
Vz/FNNC0174-0833: The apparent volume of distribution of NNC0174-0833 in the terminal phase | From pre-dose (Day 1) to Visit 7 (Day 36)
  measured in L
Change in body weight | From pre-dose (Day 1) to Visit 7 (Day 36)
  measured in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com